CLINICAL TRIAL: NCT07256054
Title: Effect of Adding High-power Pain Threshold Ultrasound to Vibration Massage on Calf Muscle Tightness in Knee Osteoarthritis Patients
Brief Title: High-power Pain Threshold Ultrasound and Vibration Massage in Treatment Knee Osteoarthritis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Doaa Rafat, Assistant professor pf physical therapy, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pt.Rec/2025-0065
Record Dates: First submitted 2025-11-15; First posted 2025-12-01 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Knee Osteoarthritis
Keywords: High-power pain threshold ultrasound; Vibration massag; Calf muscle tightness; Knee osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group (A) (Active Comparator): Group (A) received conventional treatment.
  Interventions: Other: Conventional treatment
- Group (B) (Experimental): Group (B) received conventional treatment plus vibration massage
  Interventions: Other: Conventional treatment; Other: Vibration massage
- Group (C) (Experimental): Group (C) received conventional treatment, vibration massage and the high-power pain threshold ultrasound
  Interventions: Other: Conventional treatment; Other: Vibration massage; Other: High-power pain threshold ultrasound

INTERVENTIONS:
Other: Conventional treatment — 1. TENS: Conventional TENS was used for 20 minutes to deliver asymmetrical rectangular biphasic pulsed electrical currents at a pulse repetition frequency (rate) of 100 Hz and pulse duration (width) of 250 Ksecs. The TENS was administered using two channels and four electrodes with the negative electrode (cathode) placed on the MTrP of the calf muscle and the positive electrode placed on the insertion of the muscle
  2. Calf and hamstring stretching
  3. Strengthening of the lower limb musculature (quadriceps) multi angle isometric exercises
  4. Straight leg raising exercise
  5. Mini squats
  6. Hip extension exercise
  7. Hip abduction and adduction with weights (side lying) using ankle weights
Other: Vibration massage — 1- Application of Vibration massage: Typical starting point is 30 seconds at a moderate speed for a typical trigger point (60 for chronic deep trigger points). There may be multiple trigger points in an area, each needing an application of massage. The medial gastrocnemius muscle was the focus of the first 2.5 minutes of the massage treatment, while the lateral gastrocnemius muscle was the focus of the second 2.5 minutes.
  Within 20 seconds, the massage system was shifted longitudinally in a straight line from distal to proximal and back to distal, starting at the very medial side of the treated muscle,we shifted the vibration massage unit laterally and longitudinally from distal to proximal and back to distal at the distal end of the muscle. The massage began on the medial side and ended on the lateral side for each muscle. We attempted to apply the same amount of force to the skin. The duration of the continuous vibratory massage intervention for calf muscle was 5 min (10 min )
  Arms: Group (B); Group (C)
Other: High-power pain threshold ultrasound — Application of High-power pain threshold ultrasound:
  Patient position: the subject lying down prone with foot out of bed. Therapist position: The therapist was standing at the patient's affected side's foot end.
  The high-power pain threshold ultrasound (HPPTUS) technique which US is applied in continuous mode with intensity from 0.5 to 2 watt/cm to elicit pain threshold the US probe was kept motionless, and the intensity progressively increased until the maximum level of pain patient can endure was selected, it was maintained on this level for 3 to 4 seconds and then decreased to half intensity for 15 seconds the treatment process was repeated three times
  Arms: Group (C)

SUMMARY:
Calf muscle have tendency of development of trigger points that can increase pain in patients with osteoarthritis. Purpose:To investigate the effect of adding high-power pain threshold ultrasound to vibration massage on calf muscle tightness, pain intensity, pain threshold, and knee function in knee osteoarthritis patients. Subject and methods: Sixty male and female patients diagnosed clinically by physician as having knee osteoarthritis grades II-III participated in the study. Their age ranged from 40 to 60 years. They were assigned randomly into three groups (A, B, C) equal in number. Group (A) received conventional treatment. Group (B) received conventional treatment plus vibration. Group (C) received conventional treatment, vibration and the high-power pain threshold ultrasound. Outcome measurements were taken before and after intervention, so patients received intervention for 12 sessions (three sessions per week). Tape measurement was used to measure the calf muscle flexibility, VAS to measure pain intensity, pressure algometer to measure pain threshold and WOMAC questionnaire to measure the knee functions.

DETAILED DESCRIPTION:
The current study was conducted to investigate the therapeutic effect of adding high-power pain threshold ultrasound to vibration massage on calf muscle tightness,pain intensity, pain threshold and knee function in patients with knee osteoarthritis.The study was conducted on 60 volunteer patients (age 40-60 years) suffering from unilateral knee OA grade II-III.Group (A): consisted of 20 patientsreceived the conventional physical therapy program only (Control group). Group (B): consisted of 20 patientsReceived conventional physical therapy program in addition to vibration massage. Group (C): consisted of 20 patientsreceived high-power pain threshold ultrasound in addition to conventional physical therapy program and the vibration massage. Tape measurement was used to measure the calf muscle flexibility, VAS to measure pain intensity, pressure algometer to measure pain threshold and WOMAC questionnaire to measure the knee functions. SPSS software version 22 was used to conduct all statistical analyses.

ELIGIBILITY:
Inclusion Criteria:

1. Age from 40 to 60 years' patients of chronic knee OA
2. Patient with unilateral knee OA grade II-III Kellgren and Lawrence (K/L)
3. Patients with BMI < 30 kg/m² (not being classified as obese).
4. Patients who are able to walk with painful knee OAwithoutassistive devices.
5. Patients with knee pain intensity level at least >3 cm on a 10 cm. VAS scale in activities such as going up-and downstairs, sitting and squatting.

Exclusion Criteria:

* Radiated pain from low back pain.
* No radiographic evidence of knee OA or with mild OA (grade I according to K/L classification) or with severe OA (grade IV according to K/L classification).
* Bilateral knee OA.
* Loss of joint play in tibiofemoral and patellofemoral articulations.
* Lower extremity fracture and surgery or trauma to the knee joint.
* Neurological deficit or movement disorder related to lower limb.
* Athletes or who had been treated with physiotherapy or medications during the previous 6 weeks.
* Those who could not apply vibration and percussion stimuli.
* Those who had varicose veins.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-08-30 (Actual)

PRIMARY OUTCOMES:
Calf muscle flexibility | At enrollment and after 4 weeks of treatment
  Calf Muscle Tightness Test: the subject stands a short distance away from a wall, with one leg in front of the other. Keeping the heel of the front foot on the ground, try and bend at the knee and touch the knee to the wall. If done successfully, move further away from the wall and try again. Keep repeating this action until you are unable to touch the wall. Measure the distance from the front of the foot to the wall at the maximum distance the knee could touch the wall. Repeat the same procedure for each leg.
  Scoring: measure the maximum distance from the toe to the wall. There are no norms available for this test

SECONDARY OUTCOMES:
Pain intensity | At enrollment and after 4 weeks of treatment
  Patients were asked to rate their pain intensity level on visual analogue scale in activities such as going up-and downstairs, sitting and squatting the minimum score is 1 and the maximum score is 10 higher scores mean worse outcome.
Pain threshold level | At enrollment and after 4 weeks of treatment
  pressure pain thresholds (PPT) and temporal summation of sustained pressure pain was measured by using digital algometer. The primary outcome chosen was the PPT on the stretched calf. Constant pressure stimulation at 125% of the baseline PPT pressure (obtained at the first visit) was applied for 6 minutes. The participants rated the pain intensity continuously during the constant pressure stimulation on an electronic power of 0.81 to detect a mean difference in PPT at the stretched calf (primary outcome) of 5 kPa, which from content expert viewpoint seems relevant. Pressure pain points were measured over the calf muscle belly
Knee function Assessment | At enrollment and after 4 weeks of treatment
  Universities Osteoarthritis Index (WOMAC) was used. The patient was informed with the questionnaire sub scales and was asked to fill the physical function subscale which consists of 17 items and pain which consists of 5 items. All items were evaluated from 0 which mean nothing, 1 means slight, 2 is moderate, 3 is very, and 4 is extreme. All discussions were in Arabic language.
  The scores are summed for items in each subscale, with possible ranges as follows: pain=0-20, stiffness=0-8, physical function=0-68.A total WOMAC score is created by summing the items for all three subscales (0-96) higher scores on the WOMAC indicate worse pain, stiffness, and functional limitations

CONTACTS AND LOCATIONS:
Overall Officials: Ragia M Kamel, Study Chair — Physical Therapy faculty, Cairo University
Locations (1):
- Physical Therapy faculty, Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No